CLINICAL TRIAL: NCT04106960
Title: Quantitative Investigation of the Association Between the Social and Physical Features of the Environment and Participation for Those With Complex Mental Health Difficulties Living in Supported Accommodation
Brief Title: Quantitative Investigation of Environment and Participation
Acronym: QIEP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Queen Margaret University (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Principal Investigator, Akkara Lionel Jose, PhD Student, Queen Margaret University
Other Study IDs: QIEP01
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-09

CONDITIONS: Supported Accommodation Residents; Schizophrenia, Shizotypal and Delusional Disorders; Mood Affective Disorders; Disorders of Adult Personality and Behavior
MeSH Terms: conditions — Schizophrenia; Schizophrenia, Paranoid; Mood Disorders; Behavior

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intevention Used — N/A as in the study does not have intervention in place. It is exploring the relationships between the social and physical features of the environment and participation through using standardized outcome measures.

SUMMARY:
Supported accommodation provides individuals with complex mental health difficulties the opportunity to maintain a tenancy with different levels of staff support provided to develop and maintain living skills and engage in social and work activities. Physical features of the place people live, the support they receive from staff and the individuals needs all have the potential to impact on their ability to engage in activities that enable then to have increasing independence within the community.

The study will investigate the relationship between the physical and social features of supported accommodation environments and whether this facilitates or inhibits people with complex mental health difficulties' participation in everyday life, relationships, pursuing interests and work. The study will also consider whether people's needs have an effect on the relationship between the environment and their participation. The study will analyse data collected using measures of clients' levels of participation, features of the supported accommodation environment and how needs mediates this relationship.

The aim is to inform ways of working with people with complex mental health difficulties in supported accommodation that increase opportunities for participation in the activities they need, want and enjoy doing.

DETAILED DESCRIPTION:
Mental illness is one of the main causes of disability and ill-health worldwide with severe mental illness linked to a reduced life expectancy of approximately 10-25 years. Individuals with complex mental health difficulties(CMHD) are those with severe mental illness whose conditions can result in social, cognitive and functional difficulties. These individuals possess the longest years lived with a disability and represent a large proportion of those disadvantaged or discriminated economically, socially and culturally. The impact of the social, cultural and physical environment on people with CMHD frequently resulting difficulties with participation which include isolation from friends, family and relevant services and higher levels of unemployment, subsequently, this restricts their participation in everyday roles and responsibilities. The lack of social interaction and constant low expectation of success projected onto individuals with CMHD also creates a loss of personal identity and reduces their ability to engage in activities they find meaningful. Therefore the relationship between the environment and an individual with CMHD's can be considered as dynamic, with the opportunity to participate in daily life, roles and responsibilities either being supported or restricted by the social, cultural and physical environment the person lives in.

Participation in activities that are meaningful to people with CMHD also enable them to meet their needs. Mental health needs include broad domains of health and social functioning which are essential to living and succeeding in the community. People with CMHD identify needs in relation to reframing their illness experience so they can do everyday things, having stable housing and a choice about where they live, having the ability to develop friendships, get married, earn money and have an increased sense of purpose or meaning to their day. Effectively identifying and addressing people with CMHD's needs has been linked to individual feelings of satisfaction and competence, motivation increased independence and having a greater quality of life. This introduces a link between participation and achievement of the health and social care needs of an individual where achievement of needs has been linked to increased participation in meaningful activities and improved social and emotional wellbeing.

A significant number of individuals with CMHD live in supported accommodation which aims to meet their needs and facilitate participation in daily living, social and work activities. Supported accommodation was originally developed as a result of deinstitutionalisation, which focused on moving individuals with CMHD out of hospital to live back in the community. Supported accommodation provides individuals with CMHD the opportunity to maintain a tenancy with different levels of staff support provided to develop and maintain living skills and engage in social and work activities. There is some evidence that the physical features of the place people live, and the objects or things that people require to participate in daily life and social features including the support they receive from support staff and family members have an impact on people with CMHD's opportunities to participate in activities that enable them to have increasing independence within the community. There is therefore evidence that the needs of individuals with CMHDs are associated with their level of participation in activities which in turn is influenced by environmental factors within supported accommodation. However, there is limited research available to confirm the relationship between the physical and social features of the environment and participation and the mediating effect of needs for people with CMHD living in supported accommodation.

The research will focus on identifying the relationships between environment and participation and if needs mediates this relationship within two types of supported accommodation;

1. Supported housing: tenancies in shared living with staff based on-site up to 24 hours a day. The focus is on rehabilitation, with people with CMHD supported to gain independent living skills.
2. Floating outreach services: provide support to people with CMHD living in their own self-contained tenancy. Staff are based off-site and visit individuals several times a week dependant on level of support required.

The research will use measures of the social and physical features of the supported accommodation environment, individuals' participation and need to identify the relationship between the environment and participation.

It is anticipated that the results will inform interventions for people with CMHD living in supported accommodation to maximise opportunities for participation.

Research Questions

* What is the relationship between the social and physical features of the environment and participation for people with complex mental health difficulties living in supported accommodation?
* Do needs mediate the relationship between environment and participation for people with complex mental health difficulties living in supported accommodation
* Establish the relationship between subdomains of the environment on participation for people with complex mental health difficulties living in supported accommodation.

Recruitment and Informed Consent

The detailed process is explained within the consent flowchart attached separately. The researcher will meet with staff and service managers to provide information regarding the study. They will then be asked to speak with clients about the research and provide them with the written information. A week later, the researcher will contact the service managers to confirm:

* How many clients are interested in participating in the study.
* If any clients have an attorney/welfare guardian/next of Kin that are able to consent for the research.
* A time that is convenient to meet potential participants and speak with attorney/welfare guardians.

Information on the study will be provided to the service manager for the supported accommodation, this will include participant information sheets. Clients will be approached by the service manager or support worker who will inform the researcher of clients who are willing to participate.

This will be followed by a decision making capacity process (explained in capacity flowchart attached) and gaining of consent from clients, staff and clients family members (if applicable). This will include the use of the UBACC for clients without welfare guardians/attorneys in order to determine research decision making capacity. Dependant the assessment clients will be appropriately recruited, consent forms signed and times to complete measures arranged (as seen in flowchart). The researcher will then proceed to arrange dates and times with all involved and conduct the measure tools detailed below. Interviews will be conducted within the supportive accommodation. These tools were picked in order to appropriately explore elements of the environment, needs and participation.

The study design aims to assess the environment, needs and participation through consideration of several perspectives including both staff and clients, this ensures an objective approach while also enabling the researcher to highlight any discrepancies in views as identified within the scientific justification.

Data collection and use of the measure tools will also follow theoretically proven and tested guidance that were developed for each tool. The data collection will be completed over a period of approximately one year. Throughout the process the study design takes into consideration possible complications with working with this client group with examples of this being appropriately adjusting interview styles (without moving from the base guidance of each tool) and times according to client needs.

Sample Size The study participants are the, approximately, 235 clients who are currently resident in the two types of, EHSCP managed, supported accommodation in Edinburgh; (117 clients receiving floating outreach services and 118 clients in 36 supported housing properties). Regarding the possible recruitment rate; Patel et al. conducted a large cross-sectional study assessing the proportion of individuals with psychosis willing to take part in research of 65%. Given that this is a similar population to our research study and anticipating that the 235 invited clients meet the inclusion criteria with this recruitment rate will yield approximately 153 participants.

The modelling process would initially undertake univariable regressions to identify those significant environment variables with participation prior to taking them on to the multivariable model stage. It is expected that both the univariable and multicollinearity checks will reduce the number of variables in the multivariable models. With the above recruitment figure and following Schmidt's recommendation for 15-20 subjects per variable for multivariable linear regression analysis, this would allow a model to include approximately 8-10 independent variables.

In addition bootstrapped regression estimates in the multivariable will be reported with their associated 95% confidence interval.

Proposed Analyses Descriptive statistics for the sample (e.g. age, gender, employment, diagnosis and hours of support) in the cross-sectional study will be reported with percentages and frequencies and, mean and standard deviation or median and inter-quartile range as appropriate.

To address the primary research question a regression analysis approach will be used to assess the relationships of Participation (overall score) with Environment (overall score) and Needs (figure 1 in attached documents). As the REIS is accommodation specific it will therefore be common to those participants within the same shared accommodation, and the analysis will take this in to account. Similarly for the secondary research question: an assessment of the mediating role of Needs in the relationship between Environment on Participation thereby determining the direct and indirect effects of Environment on Participation .

For the other secondary questions following the establishing of an association with environment on participation, a series of subsequent analyses will explore the impact of the environment's sub-domains on participation(overall score) and its sub-domains. Multi-collinearity will be assessed in all models.

The associated bootstrapped model regression coefficients will be reported with their 95% confidence interval.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 16 years
* English-speaking clients
* Clients with diagnoses in the following ICD-10 categories

  * F20-29 (Schizophrenia, schizotypal and delusional disorders)
  * F30-39 (Mood affective disorders)
  * F60-69 (Disorders of adult personality and behaviour)
* Clients currently residing in one of the following types of supported accommodation

  * Supported housing
  * Floating outreach services

Exclusion Criteria:

* Primary diagnosis of learning disability as identified by staff members
* Clients who are currently experiencing acute phase of illness as advised by service manager or receiving treatment from the Intensive Home Treatment Team

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The site is supported accommodation commissioned by the Edinburgh Health and Social Care Partnership (EHSCP) in Edinbrugh. The researcher will recruit participants living in two types, supported housing and floating outreach services. This is approximately 235 individuals. It is recognised that people who are resident in supported accommodation services are those with the most complex difficulties as a result of their severe mental illness. It is likely that some of the people resident in supported accommodation services will be subject to Community Compulsory Treatment Orders (CCTO) with a smaller number also having their needs managed by the Adults with Incapacity(Scotland) Act 2000.
Sampling Method: Non-Probability Sample
Enrollment: 235 (Estimated)
Dates: Start 2020-01-17 (Estimated); Primary Completion 2020-12-24 (Estimated); Study Completion 2020-12-24 (Estimated)

PRIMARY OUTCOMES:
Model of Human Occupation Screening Tool | Assessment is an interview that takes approximately 45 minutes.
  Measure of level of Participation. Participation is measured through 6 domains of Motivation for Occupation, Pattern of Occupation, Communication and interaction skills, Process skills, Motor skills and Environment. Each domain consists of 4 sub-domains whose scores will be combined. For the purpose of this study the researcher will exclude the environment domain as this would be measured by the REIS mentioned below. The domains are rated on a 4-point scale of F, A, I, R where they stands for Facilitates occupational participation, Allows occupational participation, Inhibits participation and Restricts occupational participation. Dependant on the regression model, the researcher will use both combined total scores as well as scores of specific domains and sub-domains.
Residential Environment Impact Scale | Assessment is done through three stages: a walk-around the property (15 minutes), interview with staff/staff group (30-40 minutes), interview with clients (20-45 minutes).
  Measure to assess the Environment and built for supportive environments. The REIS consists of 4 domains of Everyday Space, Everyday Objects, Enabling relationships and Structure of Activities; each domain possesses 5 sub-domains. It consists of a 4-point ordinal scale of 1,2,3,4 where 1 refers to the Environment STRONGLY INTERFERES with people's sense of identity & competence by NOT PROVIDING OPPORTUNITIES, resources, demands and constraints to engage in meaningful culturally appropriate activities. Similarly 2 stands for Interferes with by providing limited opportunity, 3 stands for supports by providing opportunities and 4 stands for strongly supports by providing exceptional opportunities. Dependant on the regression model, the researcher will use both combined total scores as well as scores of specific domains and sub-domains.

SECONDARY OUTCOMES:
Camberwell Assessment of Need Short Appraisal Scale | Interviews take approximately 30 minutes.
  Measure used to identify health and social care needs. The CANSAS is a document consisting of 22-questions assessing various health and social care needs and identifies whether a client identifies this as a need and whether this need is met or unmet. The rating scale consists of 0,1,2 and 9 where 0 is no problem with the need, 1 is met need, 2 unmet need and 9 is not known. The scoring consists of calculating the 1s and 2s separately and the total score of 1s and 2s. Due to met being the opposite of unmet, the researcher will be recording scores as a fraction of met (1s) to total needs (1s+2s).

CONTACTS AND LOCATIONS:
Overall Officials: Kirsty Forsyth, Prof, Principal Investigator — Queen Margaret University
Locations (1):
- Edinburgh Health And Social Care Partnership, Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: No
N/A no identifiable information will be published or shared.

REFERENCES:
- [Background] Whiteford HA, Degenhardt L, Rehm J, Baxter AJ, Ferrari AJ, Erskine HE, Charlson FJ, Norman RE, Flaxman AD, Johns N, Burstein R, Murray CJ, Vos T. Global burden of disease attributable to mental and substance use disorders: findings from the Global Burden of Disease Study 2010. Lancet. 2013 Nov 9;382(9904):1575-86. doi: 10.1016/S0140-6736(13)61611-6. Epub 2013 Aug 29. PMID 23993280
- [Background] WORLD HEALTH ORGANISATION (WHO), 2016. Excess mortality in persons with severe mental disorders. s.l.:World Health Organization.
- [Background] Killaspy H. Supported accommodation for people with mental health problems. World Psychiatry. 2016 Feb;15(1):74-5. doi: 10.1002/wps.20278. No abstract available. PMID 26833612
- [Background] Johnstone MJ. Stigma, social justice and the rights of the mentally ill: challenging the status quo. Aust N Z J Ment Health Nurs. 2001 Dec;10(4):200-9. doi: 10.1046/j.1440-0979.2001.00212.x. PMID 11703270
- [Background] Bastiampillai T, Allison S, O'Reilly R, Licinio J, Sharfstein SS. Can deinstitutionalisation contribute to exclusion? Lancet. 2018 Jun 2;391(10136):2210. doi: 10.1016/S0140-6736(18)30779-7. Epub 2018 Jun 1. No abstract available. PMID 29893219
- [Background] MENTAL HEALTH FOUNDATION, 2016. Fundamental Facts About Mental Health 2016, London: s.n.
- [Background] HITCH, D., PEPIN, G. & STAGNITTI, K., 2013. Engagement in Activities and Occupations by People Who Have Experienced Psychosis: A Metasynthesis of Lived Experience. British Journal of Occupational Therapy, 15 2, 76(2), pp. 77-86.
- [Background] Bejerholm U, Eklund M. Occupational engagement in persons with schizophrenia: relationships to self-related variables, psychopathology, and quality of life. Am J Occup Ther. 2007 Jan-Feb;61(1):21-32. doi: 10.5014/ajot.61.1.21. PMID 17302102
- [Background] Prior S, Maciver D, Forsyth K, Walsh M, Meiklejohn A, Irvine L. Readiness for employment: perceptions of mental health service users. Community Ment Health J. 2013 Dec;49(6):658-67. doi: 10.1007/s10597-012-9576-0. Epub 2013 Jan 19. PMID 23334300
- [Background] Mallinson T, Hammel J. Measurement of participation: intersecting person, task, and environment. Arch Phys Med Rehabil. 2010 Sep;91(9 Suppl):S29-33. doi: 10.1016/j.apmr.2010.04.027. PMID 20801276
- [Background] Priebe S, Saidi M, Want A, Mangalore R, Knapp M. Housing services for people with mental disorders in England: patient characteristics, care provision and costs. Soc Psychiatry Psychiatr Epidemiol. 2009 Oct;44(10):805-14. doi: 10.1007/s00127-009-0001-0. Epub 2009 Mar 7. PMID 19277440
- [Background] Slade M, Phelan M, Thornicroft G, Parkman S. The Camberwell Assessment of Need (CAN): comparison of assessments by staff and patients of the needs of the severely mentally ill. Soc Psychiatry Psychiatr Epidemiol. 1996 Jun;31(3-4):109-13. doi: 10.1007/BF00785756. PMID 8766455
- [Background] Piat M, Boyer R, Fleury MJ, Lesage A, O'Connell M, Sabetti J. Resident and proprietor perspectives on a recovery orientation in community-based housing. Psychiatr Rehabil J. 2015 Mar;38(1):88-95. doi: 10.1037/prj0000104. Epub 2015 Jan 5. PMID 25559078
- [Background] NELSON, D. L. & JEPSON-THOMAS, J., 2003. Occupational Form, Occupational Performance, and a Conceptual Framework for Theraputic Performance | University of Salford. In: Perspectives in human occupation: participation in life. London,Philadelphia,Pa: Lippincott Williams & Wilkins, pp. 87-155.
- [Background] Persson E, Anderberg P, Ekwall AK. A room of one's own--Being cared for in a hospital with a single-bed room design. Scand J Caring Sci. 2015 Jun;29(2):340-6. doi: 10.1111/scs.12168. Epub 2014 Sep 12. PMID 25213674
- [Background] Dunn EC, Wewiorski NJ, Rogers ES. The meaning and importance of employment to people in recovery from serious mental illness: results of a qualitative study. Psychiatr Rehabil J. 2008 Summer;32(1):59-62. doi: 10.2975/32.1.2008.59.62. PMID 18614451
- [Background] Lambri M, Chakraborty A, Leavey G, King M. Quality of life and unmet need in people with psychosis in the London Borough of Haringey, UK. ScientificWorldJournal. 2012;2012:836067. doi: 10.1100/2012/836067. Epub 2012 Nov 19. PMID 23213300
- [Background] Sheldon KM, Elliot AJ, Kim Y, Kasser T. What is satisfying about satisfying events? Testing 10 candidate psychological needs. J Pers Soc Psychol. 2001 Feb;80(2):325-39. doi: 10.1037/0022-3514.80.2.325. PMID 11220449
- [Background] Stobbe J, Wierdsma AI, Kok RM, Kroon H, Depla M, Mulder CL. Decrease in unmet needs contributes to improved motivation for treatment in elderly patients with severe mental illness. Soc Psychiatry Psychiatr Epidemiol. 2015 Jan;50(1):125-32. doi: 10.1007/s00127-014-0918-9. Epub 2014 Jul 2. PMID 24985314
- [Background] Parkinson S, Chester A, Cratchley S, Rowbottom J. Application of the Model of Human Occupation Screening Tool (MOHOST Assessment) in an Acute Psychiatric Setting. Occup Ther Health Care. 2008;22(2-3):63-75. doi: 10.1080/07380570801989465. PMID 23941373
- [Background] FISHER, G., FORSYTH, K., HARRISON, M., ANGAROLA, R., KAYHAN, E., NOGA, P., ET AL.. 201. Residential Environment Impact Scale (REIS) Version 4.0. 4 ed. Chicago, IL: University of Illinois at Chicago.
- [Background] HAYES, A. F., 2009. Beyond Baron and Kenny: Statistical Mediation Analysis in the New Millennium. Communication Monographs, 12, 76(4), pp. 408-420.
- [Background] de Heer-Wunderink C, Visser E, Caro-Nienhuis A, Sytema S, Wiersma D. Supported housing and supported independent living in the Netherlands, with a comparison with England. Community Ment Health J. 2012 Jun;48(3):321-7. doi: 10.1007/s10597-011-9381-1. Epub 2011 Jan 19. PMID 21246274
- [Background] Davidson L, Arrigo BA. Managing risk and marginalizing identities: on captivity and citizenship. Introduction. Int J Offender Ther Comp Criminol. 2013 Jun;57(6):663-5. doi: 10.1177/0306624X13480635. No abstract available. PMID 23648639
- [Background] ROWLES, G. D., 2008. Place in occupational science: A life course perspective on the role of environmental context in the quest for meaning. Journal of Occupational Science, 10, 15(3), pp. 127-135.
- [Background] HOCKING, C., 2004. The relationship between objects and identity in occupational therapy: a dynamic balance of rationalism and romanticism, s.l.: Auckland University of Technology.
- [Background] SCHMIDT, F. L., 1971. The Relative Efficiency of Regression and Simple Unit Predictor Weights in Applied Differential Psychology. Educational and Psychological Measurement, 2 10, 31(3), pp. 699-714.
- [Background] Patel R, Oduola S, Callard F, Wykes T, Broadbent M, Stewart R, Craig TK, McGuire P. What proportion of patients with psychosis is willing to take part in research? A mental health electronic case register analysis. BMJ Open. 2017 Mar 9;7(3):e013113. doi: 10.1136/bmjopen-2016-013113. PMID 28279995